CLINICAL TRIAL: NCT05594732
Title: The Effects of Different Outdoor Light Exposure Modes on Retinal Blood Flow in School Students: a Randomized Controlled Trial
Brief Title: The Effects of Different Outdoor Light Exposure Modes on Retinal Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YFZXLDX20220802
Record Dates: First submitted 2022-10-01; First posted 2022-10-26 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2022-10

CONDITIONS: Myopia
Keywords: myopia; retinal blood flow; accommodative micro-fluctuation; outdoor light exposure
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: The participants were randomly divided into the following two groups:
  1. 4000Lux natural light exposure;
  2. 10000Lux natural light exposure.
Who Masked: Participant
Masking Description: The participants were randomly divided into two groups without knowing the exposing mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weak outdoor light (Experimental): 4000Lux natural light exposure
  Interventions: Behavioral: Weak outdoor light
- Strong outdoor light (Experimental): 10000Lux natural light exposure
  Interventions: Behavioral: Strong outdoor light

INTERVENTIONS:
Behavioral: Weak outdoor light — Stay and stare far on the balcony or under the tree
  Arms: Weak outdoor light
Behavioral: Strong outdoor light — Stay and stare far in the sunlight
  Arms: Strong outdoor light

SUMMARY:
In 2020, the overall myopia rate among children and adolescents in my country was 52.7%. The COVID-19 pandemic has increased students' time of indoor eye-using, and it showed that the light exposure intensity of myopic students is lower than that of non-myopia students. Studies have found that the light wave bandwidth has a significant impact on the emmetropization of the eye, and white light can promote emmetropia more than monochromatic light. It shows that outdoor exercise has a protective effect on the occurrence and development of myopia in children and adolescents, but the specific mechanism is still unclear. Retinal blood flow is sensitive to myopic stimuli, and is a short-term indicator of the relationship between light environment and myopia. This study selected retinal blood flow as the primary outcome, aiming to compare the effects of different outdoor light exposure modes on retinal blood flow after 1 hour of intense eye use, and provide clues for the prevention and control of myopia.

DETAILED DESCRIPTION:
In 2018, eight departments including the Ministry of Education jointly issued the Implementation Plan for Comprehensive Prevention and Control of Myopia in Children and Adolescents. As of 2020, the overall myopia rate among children and adolescents in my country was 52.7%. The COVID-19 pandemic has increased students' time of indoor eye-using, and it showed that the light exposure intensity of myopic students is lower than that of non-myopia students. Studies have found that the light wave bandwidth has a significant impact on the emmetropization of the eye, and white light can promote emmetropia more than monochromatic light. It shows that outdoor exercise has a protective effect on the occurrence and development of myopia in children and adolescents, but the specific mechanism is still unclear. Retinal blood flow is sensitive to myopic stimuli, and is a short-term indicator of the relationship between light environment and myopia. Also, there is a theory that reduced choroidal blood flow causes scleral hypoxia, which leads to the development of myopia. Therefore, this study selected retinal blood flow as the primary outcome, aiming to compare the effects of different outdoor light exposure modes on retinal blood flow after 1 hour of intense eye use, and provide clues for the prevention and control of myopia.

ELIGIBILITY:
Inclusion Criteria:

* School students aged from 7 to 15, regardless of sex or gender;
* Diopter between -2.0D and 3.0D, and astigmatism not exceed 0.75D;
* No organic disease and in good general condition;
* Have obtained the consent of their parents or guardians, and can cooperate.

Exclusion Criteria:

* Suffering from amblyopia, strabismus, color weakness, congenital cataract, glaucoma and other eye diseases;
* Other circumstances judged by the investigator to be unsuitable to participate in the research.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Retinal blood flow density after relaxing for 15 minutes | Exposing to sunlight for 15 minutes
  Data collected from Optovue AngioVue OCT (macular blood data collected) for the dominant eye. The duration of relaxing was recorded by a timer.

SECONDARY OUTCOMES:
Retinal blood flow density changes between relaxing for 5 and 15 minutes | Retinal blood flow density after relaxing for 5 and 15 minutes
  The difference in retinal blood flow density was calculated between 5 and 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangui He, Principal Investigator — Shanghai Eye Hospital
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirhajianmoghadam H, Pina A, Ostrin LA. Objective and Subjective Behavioral Measures in Myopic and Non-Myopic Children During the COVID-19 Pandemic. Transl Vis Sci Technol. 2021 Sep 1;10(11):4. doi: 10.1167/tvst.10.11.4. PMID 34473223
- [Background] Rucker F. Monochromatic and white light and the regulation of eye growth. Exp Eye Res. 2019 Jul;184:172-182. doi: 10.1016/j.exer.2019.04.020. Epub 2019 Apr 21. PMID 31018118
- [Background] Xiong S, Sankaridurg P, Naduvilath T, Zang J, Zou H, Zhu J, Lv M, He X, Xu X. Time spent in outdoor activities in relation to myopia prevention and control: a meta-analysis and systematic review. Acta Ophthalmol. 2017 Sep;95(6):551-566. doi: 10.1111/aos.13403. Epub 2017 Mar 2. PMID 28251836
- [Background] Liu Y, Wang L, Xu Y, Pang Z, Mu G. The influence of the choroid on the onset and development of myopia: from perspectives of choroidal thickness and blood flow. Acta Ophthalmol. 2021 Nov;99(7):730-738. doi: 10.1111/aos.14773. Epub 2021 Feb 7. PMID 33550704
- [Derived] Zhao L, Zhang B, Wang J, Yang J, Du L, Wang T, Xu X, He X, Chen J. Short-term effects of sunlight exposure on fundus blood flow perfusion in children: a randomised controlled trial. Br J Ophthalmol. 2024 Dec 17;109(1):139-145. doi: 10.1136/bjo-2024-325715. PMID 38981665